CLINICAL TRIAL: NCT04037943
Title: NUTS for the Prevention of Cardiovascular Disease in Chinese Adults : a Randomized Controlled Trial (NUTS)
Brief Title: NUTS for the Prevention of Cardiovascular Disease in Chinese Adults
Acronym: NUTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NUTS
Record Dates: First submitted 2019-01-14; First posted 2019-07-30 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Diseases; Dyslipidemias
Keywords: Alpha linolenic acid
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: This study is a three-group parallel design trial. The paralele groups will be the control group, the low-dose intervention group, and the high-dose intervention group. Eligible participants will be randomly assigned to one of the three groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study is a single-blinded trial where investigators and outcome assessors will be blinded to the groups the participants are randomized to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose group (Experimental): Low-dose group will received 30 grams of walnuts everyday during the study period of 6 months.
  Interventions: Dietary Supplement: Walnuts 30 grams
- High-dose group (Experimental): High-dose group will received 60 grams of walnuts everyday during the study period of 6 months.
  Interventions: Dietary Supplement: Walnuts 60 grams
- Control group (No Intervention): Control group will received non-edible gifts during the study period of 6 months.

INTERVENTIONS:
Dietary Supplement: Walnuts 30 grams — Roasted walnuts without salt or sugar.
  Arms: Low-dose group
Dietary Supplement: Walnuts 60 grams — Roasted walnuts without salt or sugar.
  Arms: High-dose group

SUMMARY:
This study evaluates the feasibility of walnuts supplementation among population of high CVD risks over a period of 6 months. 70 participants will be controls receiving non-edible gifts. 70 participants will be given 30 grams of walnuts everyday and 70 participants will be given 60 grams of walnuts a day.

DETAILED DESCRIPTION:
Increased consumption of nuts improves the levels of lipid risk factors associated with cardiovascular disease and consistently relates to lower risk of cardiovascular disease (CVD) in prospective cohort studies. The estimates of health effects and potential population benefits of increased consumption of nuts are based mostly on observational data and there remains considerable uncertainty about whether higher intake of nuts will actually reduce cardiovascular outcomes. To address this uncertainty will require a well-conducted, adequately powered, large-scale, randomised control trial that tests the causal relationship between nut intake and the risk of cardiovascular diseases.

We hereby designed a 6-month walnut supplementation trial in a rural area of China with high rates of CVD, to obtain data to support and help to refine the design of a future long-term large RCT testing the effect of nut supplementation on CVD risk. The main objectives of the current trial are to assess the acceptability and adherence to two different doses of walnut supplementation (30 and 60 grams per day). The exploratory objectives are to determine the effects of walnut supplementation on cardiovascular risk factors including blood lipids, fasting glucose, and body weight.

ELIGIBILITY:
Inclusion Criteria:

1. A history of CVD, defined on the basis of a prior hospitalisation for a myocardial infarction or stroke, unstable angina, coronary artery bypass graft, percutaneous coronary intervention (with or without stenting), peripheral revascularization (angioplasty or surgery), symptomatic with documented hemodynamically-significant carotid or peripheral vascular disease, or amputation secondary to vascular disease, OR
2. Male aged >60 years, or female aged>65 years, AND

With at least two of the following risk factors:

1. Type 2 diabetes requiring treatment with at least two oral anti-hyperglycaemic agents and/or insulin
2. Systolic blood pressure > 140 mmHg while on one or more antihypertensive agents
3. Current daily smoking
4. Dyslipidaemia defined as HDL-cholesterol<1.0mmol/L or LDL-cholesterol>6.0mmol/L
5. Micro or macro albuminuria

Exclusion Criteria:

1. Allergic to nuts (history of food allergy with hypersensitivity to any of the components of nuts)
2. Other serious medical condition that prevents nut consumption (e.g. digestive disease with fat intolerance)
3. Any medical condition thought to limit survival to less than 1 year
4. Difficulty with consuming nuts (e.g. dental health issues that prevent chewing walnuts)
5. Unwilling to consume nuts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Post-intervention differences in blood plasma alpha linolenic acid between groups | From baseline to 6 months
  Blood plasma alpha linolenic acid will be measured at baseline and 6 months (end of trial).

SECONDARY OUTCOMES:
Post-intervention differences in estimated dietary nuts intake from 24h dietary recall between groups | From baseline to 6 months
  Using 24 hour dietary recall to estimate dietary nuts intake at baseline and 6 months (end of trial).
Differences in adherence and acceptability of walnuts between the high and low dose groups | From 2 week, 12 weeks to 6 months
  The adherence and acceptability of the supplement walnuts assessed by questionnaires conducted in the two intervention groups.

OTHER OUTCOMES:
Post-intervention differences in plasma total triglycerides between groups | From baseline to 6 months
  Plasma total triglycerides (mg/dL) will be measured at baseline and 6 months.
Post-intervention differences in plasma total cholesterol between groups | From baseline to 6 months
  Plasma total cholesterol (mg/dL) will be measured at baseline and 6 months.
Post-intervention differences in plasma HDL- cholesterol between groups | From baseline to 6 months
  Plasma HDL- cholesterol (mg/dL) will be measured at baseline and 6 months.
Post-intervention differences in plasma LDL- cholesterol between groups | From baseline to 6 months
  Plasma LDL- cholesterol (mg/dL) will be measured at baseline and 6 months.
Post-intervention differences in blood glucose between groups | From baseline to 6 months
  Blood glucose will be measured at baseline and 6 months.
Post-intervention differences in body weight between groups | From baseline to 6 months
  All participants' body weight will be measured at baseline and 6 months (end of trial) in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Yi Zhao, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Y, Li N, Yan N, Pan XF, Li Q, Micha R, Mozaffarian D, Huffman MD, Wang Y, Neal B, Tian M, Zhao Y, Wu JHY. Protocol for a randomized controlled trial to test the acceptability and adherence to 6-months of walnut supplementation in Chinese adults at high risk of cardiovascular disease. Nutr J. 2021 Jan 6;20(1):3. doi: 10.1186/s12937-020-00660-7. PMID 33407490